CLINICAL TRIAL: NCT00310635
Title: A Phase IV, Multi-Center, Controlled Open-Label Study to Evaluate the Safety, Tolerability and Immunogenicity of a Commercially Available Meningococcal C Vaccine When Given as First, Third or Fourth Immunization to Children 32-40 Months of Age
Brief Title: Safety, Tolerability and Immunogenicity of Meningococcal C Conjugate Vaccine to Children 32 to 40 Months of Age
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: M14P1E1; Impact N° 1453
Record Dates: First submitted 2006-04-03; First posted 2006-04-04 (Estimated); Last update posted 2006-10-26 (Estimated); Status verified 2006-10

CONDITIONS: Meningococcal Infection
Keywords: Prevention of meningococcal infection
MeSH Terms: conditions — Meningococcal Infections | interventions — serogroup C meningococcal conjugate vaccine

INTERVENTIONS:
Biological: Meningococcal C conjugate vaccine

SUMMARY:
Safety, Tolerability and Immunogenicity of Meningococcal C Conjugate Vaccine to Children 32 to 40 Months of Age

ELIGIBILITY:
Inclusion Criteria:

* Healthy children

Exclusion Criteria:

* known hypersensitivity to any vaccine component
* significant acute or chronic infections requiring systemic antibiotic treatment or antiviral therapy within the past 14 days
* ascertained or suspected disease caused by N. meningitidis
* household contact with or intimate exposure to an individual with a positive culture of N. meningitidis serogroup C within the previous 60 days

Ages: 32 Months to 40 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 241
Dates: Start 2005-06

PRIMARY OUTCOMES:
Determination of memory antibody response to Neisseria meningitidis serogroup C after 2 or 3 doses of MenC vaccine given during infancy, as measured by hBCA at day 0 and day 28.

SECONDARY OUTCOMES:
Determination of antibody titers in naïve control subjects.
Determination of persistence of antibody response after either 2 or 3 doses of MenC vaccine given during infancy and one dose of MenPS A/C vaccine given at 12 months of age.
Evaluation of the safety and tolerability of a single 0.5 mL intramuscular (IM) injection of MenC Vaccine when given to children approximately three years of age.

CONTACTS AND LOCATIONS:
Overall Officials: Vaccines - Information Services, Principal Investigator — Novartis Vaccines & Diagnostics
Locations (1):
- Mainz, Kehl, Traunreut, Mühldorf am Inn, Bad Sobernheim, Bad Kreuznach, Baldham, Speyer,, Oppenheim, Kempten, Germany